CLINICAL TRIAL: NCT00004286
Title: Phase III Multicenter Double Blind Controlled Trial of Human Immune Globulin Therapy in Previously Untreated Patients With Chronic Inflammatory Demyelinating Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Vermont (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11713; UVT-535
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: demyelinating neuropathy; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Immunoglobulins

INTERVENTIONS:
Drug: immune globulin

SUMMARY:
OBJECTIVES:

I. Compare and evaluate the response to treatment with intravenous human immune globulin (IVIG) or placebo in previously untreated patients with chronic inflammatory demyelinating polyneuropathy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a double blind, randomized, controlled study. Patients receive either intravenous human immune globulin (IVIG) or placebo infused at a rate of 40 mL/hr, increasing every 30 min to a maximum of 100 mL/hr daily over 6 to 8 hours for 2 days. On day 2, infusions of IVIG or placebo are delivered at the highest dose tolerated on day 1.

On day 21, patients receive another IVIG or placebo infusion. Following day 42, patients may choose to continue infusions of IVIG every 21 days for 2 doses.

Patients not receiving additional treatment are released from study. Patients are evaluated on days 10, 21, and 43.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Chronic inflammatory demyelinating polyneuropathy (CIDP) characterized by:

Progressive or relapsing disease or chronic stable course with elevated cerebrospinal fluid protein with normal cell counts Acquired demyelination on electrophysiologic studies Segmental demyelination on nerve histology

--Patient Characteristics--

* Not pregnant No significant medical disorders

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1996-02; Study Completion 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Rup Tandan, Study Chair — University of Vermont